CLINICAL TRIAL: NCT04069338
Title: Randomized Controlled Trial Comparing the Storz Modulith SLX-F2 and Dornier Delta III Lithotripter Machines
Brief Title: Comparison of Lithotripsy Urolithiasis Machines
Acronym: CoLUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-619
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Kidney Stone; Kidney Calculi; Ureteral Calculi; Ureterolithiasis; Urolithiasis
Keywords: Lithotripsy; Extracorporeal shockwave lithotripsy
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi; Ureterolithiasis; Urolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Storz Modulith SLX-F2 (Active Comparator): Patients receive standard of care treatment for their urolithiasis using the Device Storz Modulith SLX-F2
  Interventions: Procedure: Lithotripter
- Dornier Delta III Treatment (Active Comparator): Patients receive standard of care treatment for their urolithiasis using the Dornier Delta III lithotripter
  Interventions: Procedure: Lithotripter

INTERVENTIONS:
Procedure: Lithotripter — Patients receive standard of care treatment for their urolithiasis using one of two lithotripter machines

SUMMARY:
A comparison on the outcomes of patients undergoing shockwave lithotripsy using the Storz machine versus the Dornier machine.

DETAILED DESCRIPTION:
This is a single institution, prospective randomized controlled clinical trial comparing two lithotriper machines (the Storz Modulith LX-F2 and Dornier Delta III) in patients who are undergoing shockwave lithotripsy (SWL) as the primary management of their urinary stone. Patients record pain score on day of operation and post-operative day 1, and are followed for 1 month until they receive standard of care imaging at 1 month post-operatively.

ELIGIBILITY:
Inclusion Criteria:

- Cleveland Clinic Foundation patients planned for elective SWL with a preoperative CT performed

* Age ≥ 18 years old
* Male and female patients
* Patients of all ethnic backgrounds
* Stone size 5-15mm
* Stone location: Renal or proximal ureter
* Stone density: < 1200 Hounsfield Units
* Skin to stone distance: < 12cm
* Primary treatment for a solitary stone (must be previously untreated)

Patients must be capable of giving informed consent and must be capable and willing to enroll and participate fully with the study.

Exclusion Criteria:

* Prior treatment for specified stone

  * Multiple stones on treatment side (even if only one is treated)
  * Anticoagulated or history of coagulopathy
  * Prior ureteral stent placement
  * Technical problems/impossibility of localizing the stone on the day of intervention

Patients unable to give informed consent or unwilling to enroll or participate in the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Stone free rate | Four weeks post operative
  Presence of stone on follow up imaging

SECONDARY OUTCOMES:
Fluoroscopy time | Intra-operative
  Length of fluoroscopy exposure
Treatment Time | Intra-operative
  Length of surgical procedure
Pain Scores | Four days post-operative
  Response to visual analog scale
Complication Rates | One month post-operative
  Medical complications
Secondary Interventions required | One month post-operative
  Follow up surgery

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No